CLINICAL TRIAL: NCT02696226
Title: A Pilot Study of Subclinical Leaflet Thrombosis in Bioprosthetic Aortic Valves: A Randomized Controlled Trial
Brief Title: Frequency of Reduced Leaflet Motion After Surgical Aortic Valve Replacement and Transcatheter Aortic Valve Replacement.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Douglas Johnston, MD, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 16-084
Record Dates: First submitted 2016-02-16; First posted 2016-03-02 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-07

CONDITIONS: Aortic Valve Disorder
MeSH Terms: conditions — Aortic Valve Disease | interventions — Aspirin; Clopidogrel; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SAVR Warfarin Arm (Experimental): Warfarin arm-(target INR of 2-3)
  Interventions: Drug: SAVR Warfarin
- TAVR Warfarin and Clopidogrel Arm (Experimental): Warfarin (target INR of 2-3) and Clopidogrel (75mg/day) arm
  Interventions: Drug: TAVR Warfarin and clopidogrel
- SAVR Aspirin Arm (Experimental): Aspirin arm (81mg/day)
  Interventions: Drug: SAVR Aspirin
- TAVR Aspirin and Clopidogrel Arm (Experimental): Aspirin (81mg/day) and Clopidogrel (75mg/day) arm
  Interventions: Drug: TAVR Aspirin and clopidogrel

INTERVENTIONS:
Drug: SAVR Warfarin — Warfarin treatment for 12 weeks with a target INR of 2-3 Warfarin treatment to begin on postoperative day 1-3 according to the patient's clinical status When warfarin treatment is discontinued, patients will be treated according to standard of care (aspirin 81 mg/day) indefinitely
  Other Names: Coumadiin
  Arms: SAVR Warfarin Arm
Drug: SAVR Aspirin — Aspirin (81 mg/day) to begin within 1-3 postoperative days according to the patient's clinical status and continue indefinitely per standard of care.
  Other Names: Aspirin
  Arms: SAVR Aspirin Arm
Drug: TAVR Warfarin and clopidogrel — Begin Warfarin and clopidogrel (75 mg/day) treatment within 1-3 days postop for 12 weeks with a target INR of 2-3 When warfarin is discontinued, begin aspirin (81 mg/day) and continue aspirin/clopidogrel for 12 weeks At 24 weeks, study treatment will end and patients will be treated according to standard of care (aspirin 81 mg/day) indefinitely
  Other Names: Coumadin; Plavix
  Arms: TAVR Warfarin and Clopidogrel Arm
Drug: TAVR Aspirin and clopidogrel — Aspirin (81 mg/day) and clopidogrel (75 mg/day) in periprocedural period and continue for 24 weeks At 24 weeks, study treatment will end and patients will be treated according to standard of care (aspirin 81 mg/day) indefinitely
  Other Names: Plavix
  Arms: TAVR Aspirin and Clopidogrel Arm

SUMMARY:
This is a prospective, randomized pilot study in patients undergoing Sugical Aortic Valve Replacement (SAVR) and Transcatheter Aortic Valve Replacement (TAVR) to estimate the incidence of reduced leaflet motion and assess the impact of perioperative anticoagulation on the incidence of reduced leaflet motion.

DETAILED DESCRIPTION:
This will be a pilot prospective randomized controlled trial.The study will enroll 50 adult patients scheduled to undergo SAVR and 50 adult patients scheduled to undergo TAVR. Subjects who satisfy Inclusion/Exclusion Criteria will be approached for informed consent. Those who give informed consent will be enrolled. After induction of anesthesia, a computer program will be used to randomize patients to one of the 2 treatment groups.

1. SAVR patients will get either Warfarin or aspirin
2. TAVR patients will get either Warfarin or aspirin.

Patients will be seen at 4-6 weeks postoperatively for Transthoracic ECHO (TTE), 4 dimensional (4D), Multidetector computed tomography (MDCT) scan and review of medical history. Phone follow up at 6,9 and 12 months post-operatively.

Data from this pilot study will enable us to determine the feasibility of a larger randomized controlled clinical trial to investigate the phenomenon of reduced leaflet motion/subclinical valve thrombosis and, possibly, its clinical importance

ELIGIBILITY:
Inclusion Criteria:

Scheduled for SAVR or TAVR

* Age > 18 years
* Able and willing to give informed consent
* Able and willing to return for follow up

Exclusion Criteria:

* Contraindications to warfarin, Plavix or aspirin
* Pre-existing medical indication for warfarin, Plavix or aspirin
* History of previous cardiac surgery
* History of previous coronary artery stenting
* Requirement for concomitant coronary artery bypass grafting or mitral valve surgery or surgical treatment of an ascending aortic aneurysm
* Contraindications to contrast-enhanced MDCT including anaphylactic iodine allergy, uncontrolled atrial fibrillation, renal dysfunction (GFR < 60 ml/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Johnston, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SAVR Warfarin Arm | TAVR Warfarin and Clopidogrel Arm | SAVR Aspirin Arm | TAVR Aspirin and Clopidogrel Arm
Started | 1 | 0 | 2 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 2 | 0
Not completed — Study terminated - lack of enrollment | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated - lack of enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | SAVR Warfarin Arm | TAVR Warfarin and Clopidogrel Arm | SAVR Aspirin Arm | TAVR Aspirin and Clopidogrel Arm | Total
Number analyzed (Participants) | 1 | 0 | 2 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants] — Study was terminated - low number of participants did not allow for data analysis Population: Study terminated - lack of enrollment
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 0 | 0 | 2 | 0 | 2
    >=65 years | 1 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — Data was not analyzed due to low enrollment Population: Data was not analyzed due to low enrollment - Study terminated
  Participants
    Female | 0 | 0 | 1 | 0 | 1
    Male | 1 | 0 | 1 | 0 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Leaflet Motion
Description: Frequency of reduced leaflet motion related to perioperative anticoagulation with warfarin as measured by 4DMCT data. (<50% reduction in motion), moderately reduced (50 to 70% reduction), severely reduced (>70% reduction), or immobile (lack of motion of at least one valve leaflet).
Time Frame: 4-6 weeks post procedure
Population: Study terminated
Arm/Group | SAVR Warfarin Arm | TAVR Warfarin and Clopidogrel Arm | SAVR Aspirin Arm | TAVR Aspirin and Clopidogrel Arm
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Only 2 arms of the trial had enrollment (SAVR Warfarin / SAVR Aspirin). Adverse event information is reported only for these arms
Arm/Group | SAVR Warfarin Arm | TAVR Warfarin and Clopidogrel Arm | SAVR Aspirin Arm | TAVR Aspirin and Clopidogrel Arm
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT02696226/Prot_SAP_000.pdf